CLINICAL TRIAL: NCT04694677
Title: Safety of Tranexamic Acid Versus Misoprostol in Reducing Blood Loss in Myomectomy.
Brief Title: Safety of Tranexamic Acid in Reducing Blood Loss Myomectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Myomectomy
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women receiving tranexamic acid (Active Comparator)
  Interventions: Drug: women receiving tranexamic acid
- women receiving misoprostol (Active Comparator)
  Interventions: Drug: women receiving misoprostol

INTERVENTIONS:
Drug: women receiving tranexamic acid — women receiving tranexamic acid during myomectomy
  Arms: women receiving tranexamic acid
Drug: women receiving misoprostol — women receiving misoprostol in myomectomy
  Arms: women receiving misoprostol

SUMMARY:
Uterine leiomyomas (fibroids) are the most common benign tumors among women . Fibroids are found in approximately 15% to 30% of women in the reproductive age group

DETAILED DESCRIPTION:
Although most of them are asymptomatic, 20-50% of fibroids may cause problems such as heavy menstrual bleeding, anemia, pelvic pain, pressure symptoms from extrinsic compression of the colorectal and urinary tract, infertility, and recurrent pregnancy losses, where surgical intervention is often indicated

ELIGIBILITY:
Inclusion Criteria:

* women with myomas

Exclusion Criteria:

* with with malignant lesions

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with myomas
Enrollment: 60 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
the number of women who will have less blood loss | 48 hours
  how many women will have less blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Director — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt